CLINICAL TRIAL: NCT06279000
Title: Colchicine in Patients at Cardiac Risk Undergoing Major Non-Cardiac Surgery: Prospective, Randomized, Double-blinded, Placebo-controlled, Multi-centre Study
Brief Title: Colchicine in Patients at Cardiac Risk Undergoing Major Non-Cardiac Surgery
Acronym: COLCAT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Dr. Timur Yurttas, Principal Investigator, Senior Anaesthesiologist, Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTU 22/025
Record Dates: First submitted 2024-02-12; First posted 2024-02-26 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-09

CONDITIONS: Cardiovascular Diseases; Cardiovascular Complication; Perioperative Complication; Myocardial Injury; Myocardial Injury After Noncardiac Surgery (MINS)
Keywords: Perioperative Cardiovascular Risk; myocardial injury; major adverse cardiac events; colchicine
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: randomized, double-blinded, placebo-controlled, multicenter
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, anaesthesia providers and all other health care workers involved in the treatment and the study personal will be blinded to the group allocation by provision of equal looking study drugs (verum and placebo), which are repacked for blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Experimental): The first dose of the IMP is administered in the evening prior to the surgical procedure. Administrations of the study drug follow a 1-0-1 schedule (colchicine 0.5 mg per intake). The last study drug is administered in the evening of the third postoperative day.
  Interventions: Drug: Colchicine
- Control (Placebo) (Placebo Comparator): Patients in the control group will receive the same perioperative anaesthetic, surgical and medical treatment as patients in the experimental group, the sole difference being that patients will be given a placebo instead of the IMP colchicine.
  The first dose of the placebo is administered in the evening prior to the surgical procedure. Administrations of the placebo follow a 1-0-1 schedule. The last placebo is administered in the evening of the third postoperative day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — Colchicine Group:
  IMP = Colchicine (0.5 mg, enteral) first application in the evening before day of surgery, following a 1-0-1 regimen until the third postoperative day, ending with the application of the ninth dose. Colchicine tablets are provided as 1 mg tablets with a score, which must be divided before ingestion.
  Arms: Colchicine
Drug: Placebo — Placebo Group:
  Placebo (identical to IMP in appearance and application) first application in the evening before day of surgery, following a 1-0-1 regimen until the third postoperative day, ending with the application of the ninth dose. Placebo tablets are provided as tablets with a score, which must be divided before ingestion.
  Other Names: Control
  Arms: Control (Placebo)

SUMMARY:
Perioperative myocardial injury and major adverse cardiovascular events (MACE) are common causes of morbidity and mortality in patients at increased cardiovascular risk undergoing non-cardiac surgery.

However, research in recent years has yielded limited preventive and therapeutic measures for myocardial injury/MACE. Recent studies in patients with chronic and acute coronary artery disease have shown that colchicine administration can reduce the risk of cardiovascular events.

These encouraging results in non-surgical patients ask for a similar investigation in patients undergoing major non-cardiac surgery. The aim of the proposed study is to investigate the effects of perioperative colchicine administration on the incidence of myocardial injury/MACE.

DETAILED DESCRIPTION:
This double-blind, placebo-controlled study is conducted at the Cantonal Hospital St. Gallen and the University Hospital Basel, Switzerland. The investigators intend to expand the participant recruitment to other centers. Inclusion criteria encompass patients' cardiovascular risk profile and vascular, orthopedic, visceral, and thoracic surgical procedures with a high risk as determined by the recognized incidence of troponin dynamics. Patients are informed during preoperative consultation and provide consent prior to randomization to the colchicine or placebo groups. The preoperative assessment includes medical history, medication use and physical capacity. Baseline values and cardiac biomarkers, are determined through routine laboratory tests. Study medication is administered from the evening before surgery until the third postoperative day. Daily high-sensitivity cardiac troponin T (hs-cTnT) testing is performed until the fourth day. Visits monitor primary, secondary, and safety endpoints, with standard treatment for complications. Post-hospitalization, cardiovascular events will be recorded until postoperative day 30 and for one year post-surgery to assess long-term outcomes.

The primary objective is to evaluate the efficacy of perioperative colchicine administration in cardiac-risk patients undergoing major non-cardiac surgery, with the aim of reducing the myocardial injury incidence until postoperative day 4 and mitigate postoperative MACE until postoperative day 30. Secondary objectives include whether perioperative administration of colchicine reduces new-onset atrial fibrillation incidence postoperatively (until discharge) compared to placebo, to quantify the maximum increase in postoperative hs-cTnT concentrations until postoperative day 4 and to assess the impact of perioperative colchicine administration on long-term survival and morbidity (composite of MACE) after one year. The safety objectives are the incidence of gastrointestinal adverse events and clinically adverse events attributable to the administration of colchicine.

ELIGIBILITY:
Inclusion Criteria:

undergoing major non-cardiac surgery in general anaesthesia will be included. Major non-cardiac surgery is defined as:

* vascular surgery (with the exception of arteriovenous shunt, vein stripping procedures and carotid endarterectomies)
* intraperitoneal surgery
* intrathoracic surgery
* major orthopaedic surgery (spinal surgery or joint replacement surgery)
* at cardiovascular risk, defined as meeting at least 1 of the following 6 criteria:

  * preoperative n-terminal pro brain natriuretic peptide (NT-proBNP) ≥ 200 ng/l
  * history of coronary artery disease
  * history of peripheral vascular disease
  * history of stroke
  * undergoing major vascular surgery, with the exception of arteriovenous shunt, vein stripping procedures and carotid endarterectomies
  * fulfilment of any 3 of the 8 following criteria:

    * undergoing major surgery (intrathoracic, intraperitoneal or supra-inguinal vascular surgery)
    * any history of congestive heart failure or history of pulmonary oedema
    * anamnestic transient ischemic attack (TIA)
    * diabetes under treatment with either oral antidiabetic agent or insulin
    * age > 70 years
    * history of hypertension
    * serum creatinine > 175 mumol/l or calculated creatinine clearance < 60 ml/min/1.73m2 (cockcroft gault)
    * history of smoking within 2 years of surgery
    * planned surgical time ≥ 90 minutes
    * planned postoperative hospital stay at least 1 night

Exclusion Criteria:

* no written consent
* inclusion in other clinical trial with direct impact on perioperative medication
* previously reported side effects or reported intolerance from colchicine (e.g., allergic reaction or significant sensitivity to colchicine or an auxiliary substance of the IMP)
* pregnancy or planned pregnancy and/or breast feeding
* clinically significant history of drug or alcohol abuse within the last year
* very severe frailty (≥ 8 clinical frailty scale)
* patient with inflammatory bowel disease (e.g., Morbus Crohn or Colitis ulcerosa)
* patient taking colchicine for other indications (e.g., familial Mediterranean fever, gout)
* severe renal impairment (eGFR < 30 ml min -1 1.73 m2 -1) or end-stage renal disease with indication for haemodialysis
* history of solid organ or bone marrow transplantation
* systemic immune-suppression (medication (steroids >30mg cortisol-equivalent per day, tacrolimus etc...) or disease (e.g., myelodysplastic syndrome)
* severe hepatic impairment with history of cirrhosis
* chronic active hepatitis or functional disorders defined as alanine aminotransferase greater than three times the upper limit of normal
* anticipated post-operative administration of CYP3A4 metabolized substances like cyclosporine, ketoconazole, clarithromycin, verapamil, quinidine, diltiazem or ritonavir
* Any other condition that the investigator would consider a risk to the patient if the latter were to participate in the study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | until postoperative day 30
  Proportion of patients developing MACE in the peri- postoperative course. MACE is defined as a composite of any of the following within 30 days following surgery:
  * Acute coronary syndrome
  * New/worsening congestive heart failure
  * Coronary revascularization
  * Stroke
  * All-cause mortality
  * Cardiovascular death
Myocardial Injury | until postoperative day 4
  Proportion of patients developing myocardial injury in the peri- postoperative course. The primary outcome is a composite of myocardial injury and 30-day MACE. Myocardial injury is defined as an absolute perioperative rise in hs-cTnT of ≥ 14 ng/l above preoperative values (or between two postoperative measurements, if preoperative hs-cTnT is missing).

SECONDARY OUTCOMES:
New onset Atrial fibrillation | From beginning of surgery/surgical procedures until the date of first documented occurrence or until postoperative day 30/discharge from hospital, whatever comes first
  Proportion of patients developing new-onset atrial fibrillation in the peri- postoperative course. The time frame includes the time from beginning of surgery (ECG monitoring in the peri- and early postoperative course on postoperative care unit/intensive care unit) until the date of first documented occurrence of atrial fibrillation (perioperative monitoring by daily nurse-controlled pulse examination, verified by an ECG in case of suspected arrhythmia/atrial fibrillation). These monitoring procedures take place until the discharge from the hospital.
postoperative high sensitive cardiac Troponin T concentrations | until postoperative day 4
  Comparison of postoperative hs-cTnT concentrations (maximal increase from individual baseline & the area under the curve) until postoperative day 4 between the study groups
long term cardiovascular outcome | until 1 year after surgery
  Proportion of patients developing MACE in regard of long term cardiovascular outcome after surgery.1-year composite endpoint of MACE (composite of acute coronary syndrome, new or worsening congestive heart failure, coronary revascularization, stroke, all-cause mortality and cardiovascular mortality) as a marker of long-term postoperative outcome.

OTHER OUTCOMES:
Gastrointestinal adverse events | From the first intake of the study drug until 72 hours after the last intake of the study drug (i.e., postoperative day 6) or until discharge from the hospital, whatever comes first
  Proportion of patients developing gastrointestinal side effects as: diarrhoea, abdominal cramping, abdominal pain, vomiting, nausea after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Cantonal Hospital St. Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided